CLINICAL TRIAL: NCT00316043
Title: Prevention of Renal Failure in Children With Urinary Tract Infections in General Practice: Current Clinical Management, Possibilities for Improvement and Potential Cost-Efficiency
Brief Title: Prevention of Renal Failure in Children With Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: WOK_PNKU_01; OV02 (Dutch Kidney Foundation)
Record Dates: First submitted 2006-04-14; First posted 2006-04-19 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Urinary Tract Infections
Keywords: Urinary tract infections; Renal failure; Renal scarring; Prevention; Primary Care; General Practice; Intervention Studies; Children
MeSH Terms: conditions — Urinary Tract Infections; Renal Insufficiency | interventions — General Practitioners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Written information for parents
Behavioral: Distance learning package for General Practitioners
Behavioral: Distance learning package for practice assistants

SUMMARY:
The aim of the study is to describe the current clinical management of young children with urinary tract infections in Dutch primary care and also to describe the possibilities for improvement and potential cost-efficiency of improved care in the light of preventing renal failure.

DETAILED DESCRIPTION:
The aim of the study is to describe the current clinical management of young children with urinary tract infections in Dutch primary care and also to describe the possibilities for improvement and potential cost-efficiency of improved care in the light of preventing renal failure.

The 4 phases of the study contain the following questions:

* Phase 1: What is the current clinical management of urinary tract infections in young children in primary care?
* Phase 2: What are the possibilities for improving the clinical management of urinary tract infections and are these improvements practically achievable?
* Phase 3: What is the cost-efficiency of the several interventions for improving clinical management of urinary tract infections
* Phase 4: What is the influence of the intervention on clinical management?

ELIGIBILITY:
Inclusion Criteria:

* children between 0-12 years of age with a proven urinary tract infection in general practice

Exclusion Criteria:

-

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2006-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Number of antibiotic prescriptions | 10 days after 1st contact with GP
Number of referrals | 10 days after 1st contact with GP
Number of follow-up appointments | 10 days after 1st contact with GP

CONTACTS AND LOCATIONS:
Overall Officials: Michel Wensing, dr., Principal Investigator — UMC St Radboud
Locations (1):
- UMC St Radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Ahmed SM, Swedlund SK. Evaluation and treatment of urinary tract infections in children. Am Fam Physician. 1998 Apr 1;57(7):1573-80, 1583-4. PMID 9556646
- [Background] Owen D, Vidal-Alaball J, Mansour M, Bordeaux K, Jones KV, Edwards A. Parent's opinions on the diagnosis of children under 2 years of age with urinary tract infection. Fam Pract. 2003 Oct;20(5):531-7. doi: 10.1093/fampra/cmg507. PMID 14507794
- [Background] Harmsen, M et al. Urinary tract infections in young children: high guideline adherence of triage nurses at general practice co-operatives. Quality in Primary Care, 13: 241-7, 2005
- [Background] Kwok WY, de Kwaadsteniet MC, Harmsen M, van Suijlekom-Smit LW, Schellevis FG, van der Wouden JC. Incidence rates and management of urinary tract infections among children in Dutch general practice: results from a nation-wide registration study. BMC Pediatr. 2006 Apr 4;6:10. doi: 10.1186/1471-2431-6-10. PMID 16584577
- [Background] Jacobson SH, Eklof O, Eriksson CG, Lins LE, Tidgren B, Winberg J. Development of hypertension and uraemia after pyelonephritis in childhood: 27 year follow up. BMJ. 1989 Sep 16;299(6701):703-6. doi: 10.1136/bmj.299.6701.703. PMID 2508881
- [Background] Vernon SJ, Coulthard MG, Lambert HJ, Keir MJ, Matthews JN. New renal scarring in children who at age 3 and 4 years had had normal scans with dimercaptosuccinic acid: follow up study. BMJ. 1997 Oct 11;315(7113):905-8. doi: 10.1136/bmj.315.7113.905. PMID 9361538
- [Background] Hansson S, Bollgren I, Esbjorner E, Jakobsson B, Marild S. Urinary tract infections in children below two years of age: a quality assurance project in Sweden. The Swedish Pediatric Nephrology Association. Acta Paediatr. 1999 Mar;88(3):270-4. doi: 10.1080/08035259950170015. PMID 10229036
- [Background] Harmsen M, Wensing M, van der Wouden JC, Grol RP. Parents' awareness of and knowledge about young children's urinary tract infections. Patient Educ Couns. 2007 May;66(2):250-5. doi: 10.1016/j.pec.2006.12.009. PMID 17445745
- [Background] Harmsen M, Wensing M, Braspenning JC, Wolters RJ, van der Wouden JC, Grol RP. Management of children's urinary tract infections in Dutch family practice: a cohort study. BMC Fam Pract. 2007 Mar 13;8:9. doi: 10.1186/1471-2296-8-9. PMID 17355617
- See also: Related Info — http://www.wokresearch.nl